CLINICAL TRIAL: NCT06406166
Title: Clinical Efficacy of Lifei Xiaoji Wan in Treatment of Advanced NSCLC
Brief Title: Lifei Xiaoji Wan in Treatment of Advanced NSCLC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCM for advanced NSCLC
Record Dates: First submitted 2024-04-16; First posted 2024-05-09 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-05

CONDITIONS: Advanced Non Small Cell Lung Cancer
Keywords: advanced non small cell lung cancer; traditional Chinese medicine; randomized controlled trial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trial group (Experimental): The patients in the trial group received routine Western medicine treatments, and oral Lifei Xiaoji Wan (10 pills/time, 3 times/day).
  Interventions: Drug: Lifei Xiaoji Wan; Other: Conventional treatment with Western medicine
- control group (No Intervention): The patients in the control group received routine Western medicine treatments.

INTERVENTIONS:
Drug: Lifei Xiaoji Wan — The Lifei Xiaoji Wan consists of ginseng, blackhead, rhubarb, aster, forehu, and thin on
  Arms: trial group
Other: Conventional treatment with Western medicine — Conventional treatment with Western medicine
  Arms: trial group

SUMMARY:
This study is to evaluate the clinical efficacy of Lifei Xiaoji Wan for advanced non-small cell lung cancer (NSCLC), establish the treatment scheme, and obtain high-quality clinical evidence.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) is a disease with high morbidity and mortality, poor prognosis, and a lack of safe and effective treatment. Lifei Xiaoji Wan has significant advantages in the treatment of advanced NSCLC, but the a lack of high-level clinical evaluation evidence and accurate mechanism of action research. According to the previous animal experiments of the team, it was proved that Lifei Xiaoji Wan can significantly inhibit the tumor growth ability of lung cancer mice, and inhibit the proliferation, clonal formation, and migration ability of lung cancer cells. This topic intends to adopt the method of multicenter randomized controlled study to observe the Lifei Xiaoji Wan for advanced NSCLC patients' overall survival (OS), progression-free survival (PFS), Functional Assessment of Cancer Therapy-Lung (FACT-L), TCM symptoms and syndrome and safety, help to clarify the role of Lifei Xiaoji Wan in TCM prevention and treatment of lung cancer, can provide high-level evidence for TCM prevention and treatment of lung cancer research and clinical.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of NSCLC.
2. The tumor stage (TNM) stage is from III to IV.
3. 18-80 years old.
4. The expected survival period is> 3 months.

Exclusion Criteria:

1. Early-stage patients with prior surgery and no recurrence.
2. Patients with serious dysfunction of the heart, liver, heart, kidney, and other important organs.
3. Mental illness and other patients were unable to complete the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year.
  Time from enrollment to patient death.
Progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year.
  Time from enrollment to objective tumor progression or all-cause death.

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy-Lung (FACT-L) | Change from baseline the scores of FACT-L at month 2, 4, 6, 8, 10 and 12.
  Including the physiological status, social / family status, emotional status, functional status and additional concerns, with a total score of 0-144. The higher the score, the more severe the symptoms will be.
TCM symptoms and syndrome | Change from baseline the TCM symptoms and syndrome at month 2, 4, 6, 8, 10 and 12.
  The improvement of the clinical symptoms, such as cough, expectoration, chest tightness, shortness of breath, fatigue, weakness, and loss of appetite.
Response Evaluation Criteria in Solid Tumours (RECIST) | Change from baseline the RECIST at month 2, 4, 6, 8, 10 and 12.
  patients were collected on Computed Tomography (CT) for imaging analysis and measurement, to observe the changes of tumor bodies and lesions, and to evaluate the efficacy on tumor.
Tumor markers CEA | Change from baseline the levels of tumor markers at month 2, 4, 6, 8, 10 and 12.
  Peripheral blood of patients was collected to observe the changes of CEA.
Tumor markers CA211 | Change from baseline the levels of safety indicators at month 2, 4, 6, 8, 10 and 12.
  Peripheral blood of patients was collected to observe the changes of CA211.
Tumor markers Squamous Cell Careinoma Antigen | Change from baseline the levels of safety indicators at month 2, 4, 6, 8, 10 and 12.
  Peripheral blood of patients was collected to observe the changes of Squamous Cell Careinoma Antigen.
Complete blood count: White blood cells levels | Change from baseline the levels of white blood cells at month 2, 4, 6, 8, 10 and 12.
  white blood cells levels
Complete blood count: Haemoglobin levels | Change from baseline the levels of levels at month 2, 4, 6, 8, 10 and 12.
  haemoglobin levels
Complete blood count: Platelet levels | Change from baseline the levels of Platelet at month 2, 4, 6, 8, 10 and 12.
  Platelet levels
Liver function: ALT levels | Change from baseline the levels of ALT at month 2, 4, 6, 8, 10 and 12.
  ALT levels
Liver function: AST levels | Change from baseline the levels of AST at month 2, 4, 6, 8, 10 and 12.
  AST levels
Renal function: BUN levels | Change from baseline the levels of BUN at month 2, 4, 6, 8, 10 and 12.
  BUN levels
Renal function: Cr levels | Change from baseline the levels of Cr at month 2, 4, 6, 8, 10 and 12.
  Cr levels

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No